CLINICAL TRIAL: NCT03593421
Title: Phase II, Open Label Adaptive Design Dose Finding Study to Investigate Effect of Synthetic PreImplantation Factor (sPIF) in Patients With High Panel Reactive Antibodies
Brief Title: Phase 2 Dose Finding sPIF in Patients With High Panel Reactive Antibodies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: BioInceptdecided not to pursue this drug target at this time.
Sponsor: Christopher O'Brien, MD (Other)
Collaborators: BioIncept LLC (Industry)
Responsible Party: Sponsor-Investigator, Christopher O'Brien, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20171060; sPIF-US-PRA-001 (Other: University of Miami)
Record Dates: First submitted 2018-06-07; First posted 2018-07-20 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Panel Reactive Antibodies
MeSH Terms: interventions — preimplantation factor, synthetic

STUDY DESIGN:
Intervention Model Description: open label, adaptive design, dose finding study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- synthetic preImplantation factor 1 mg/kg (Experimental): Patients will be dosed SQ with 14 doses of sPIF
  Interventions: Drug: synthetic PreImplantation Factor
- synthetic preImplantation factor 2 mg/kg (Experimental): Patients will be dosed SQ with 14 doses of sPIF
  Interventions: Drug: synthetic PreImplantation Factor
- synthetic preImplantation factor 3 mg/kg (Experimental): Patients will be dosed SQ 14 doses
  Interventions: Drug: synthetic PreImplantation Factor
- synthetic preImplantation factor 4 mg/kg (Experimental): Patients will be dosed SQ with 14 doses of sPIF
  Interventions: Drug: synthetic PreImplantation Factor
- synthetic preImplantation factor 5 mg/kg (Experimental): Patients will be dosed SQ with 14 doses of sPIF
  Interventions: Drug: synthetic PreImplantation Factor

INTERVENTIONS:
Drug: synthetic PreImplantation Factor — peptide
  Other Names: sPIF

SUMMARY:
This is an open labeled dose finding adaptive design study. Patients with elevated cPRA values, 30-60% will be recruited and administered sPIF injected subcutaneously for 14 doses; one dose on Monday, Wednesday, Friday, or Tuesday, Thursday, Saturday, per individual patient dialysis schedule.

DETAILED DESCRIPTION:
The purpose of this study is to determine the sPIF dose that reduces serum cPRA to <30%, when administered 14 doses. Safety, tolerability, and efficacy will be evaluated at day 42 and and day 84. The suitability of a patient to receive a kidney transplant will also be monitored up to 6 months after Day 84. Safety and tolerability will be assessed at each of the increased doses and throughout the treatment duration. Exploratory analysis of blood indices will be carried out and changes based on history, physical and laboratory exams will be assessed according to the 12 systems.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient male and females 18-75 years old
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Calculated panel reactive antibody (cPRA) >30% and <60% with a threshold using mean fluorescent intensity (MFI) of 3,000 or standard fluorescence intensity (SFI) of 60,000 over six months.
* Women who are of childbearing potential must have a negative serum pregnancy test prior to being enrolled in the study and agree to use effective method of contraception throughout the 84-day study.
* Patients on kidney dialysis 3.3 Exclusion Criteria
* Patients not capable of following through the treatment for various reasons as determined by treating physicians
* Pregnant females
* Requiring blood transfusions
* Have an active infection
* Infection with hepatitis C virus (HCV) or hepatitis B virus(HBV) or human immunodeficiency virus (HIV), lack of documentation of treatment of a positive PPD, baseline leukopenia, white blood cell count (WBC) <4.0, thrombocytopenia (platelet count <100,000/mm) or difficult to treat anemia, a hematocrit chronically <25% on intravenous iron and EPO (erythropoietin) therapy
* Active cancer within 5 years
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of multiple ascending, subcutaneously administered doses of sPIF in patients with high panel reactive antibodies (PRA) with no SAEs greater than grade 3 | 84 days
  No grade SAE > Grade 3
Evaluate the pharmacokinetics of sPIF levels in the circulation after multiple ascending, subcutaneously administered doses of sPIF by measurement of sPIF in circulation | 84 days
  sPIF circulating levels are assessed following dialysis and post-first injection at 1, 2, and 4 hours and before last sPIF dose, trough values.
Evaluate the effect of sPIF on serum cPRA following administration of multiple ascending, subcutaneously administered doses as determined by CPRA levels | 84 days
  Determine cPRA levels

SECONDARY OUTCOMES:
Determine the percentage of patients in remission ass determined by CPRA less than 30% | 84 days
  Determine cPRA levels as defined by <30% until day 42, and sustained until day 84. Analysis is based on decrease in cPRA percent, median fluorescent intensity (MFI) and standard fluorescent intensity (SFI) analysis.
Assess number of patients receiving a kidney transplant within 6 months post-day 84 as dertermined by patients being available for kidney transplant | 6 months post study drug treatment
  Determine number of patients eligible for kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: eytan barnea, MD, Principal Investigator — BioIncept LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnea ER, Rambaldi M, Paidas MJ, Mecacci F. Reproduction and autoimmune disease: important translational implications from embryo-maternal interaction. Immunotherapy. 2013 Jul;5(7):769-80. doi: 10.2217/imt.13.59. PMID 23829627